CLINICAL TRIAL: NCT02462707
Title: Phase 1 Study Of Pf-03084014 To Evaluate Safety And Pharmacokinetics In Japanese Patients With Advanced Solid Tumors
Brief Title: A Study Of PF-03084014 In Japanese Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8641021
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-03084014 (Experimental)
  Interventions: Drug: PF-03084014

INTERVENTIONS:
Drug: PF-03084014 — gamma-secretase inhibitor, formulated in tablets for oral administration containing 10 mg, 50 mg and 100 mg. Patient will receive 80 mg, 100 mg or 150 mg twice daily of PF-03084014 with continuous dosing schedule

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose for PF-03084014 single-agent administration in Japanese patients with advanced solid tumors. Pharmacokinetics and the overall safety profile of PF-03084014 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced solid tumors that is resistant to standard therapy or for which no standard therapy is available.
* Age ≥18 years.
* ECOG Performance Status (PS) must be 0 or 1.
* Adequate Bone Marrow Function
* Adequate Renal Function
* Adequate Liver Function
* Resolved acute effects of any prior therapy to baseline severity or Grade ≤1

Exclusion Criteria:

* Patients with known brain metastases
* Major surgery within 4 weeks of starting study treatment
* Radiation therapy within 2 weeks of starting study treatment
* Systemic anti cancer therapy within 2 weeks (4 weeks for antibody) of starting study treatment
* Previous high dose chemotherapy requiring stem cell rescue
* Prior irradiation to >25% of the bone marrow
* Prior treatment with a Notch signal inhibitor
* Known malabsorption syndrome or other condition that may impair absorption of study medication
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism
* Current use or anticipated need for known strong and/or moderate CYP3A4 inhibitors
* Current use or anticipated need for known strong CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
First-cycle Dose Limiting Toxicities | during the first 28 days from the first dose

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
QTc interval | from the first dose to the last dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Apparent Oral Clearance (CL/F) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Apparent Volume of Distribution at steady state (Vss/F) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Minimum Observed Plasma Trough Concentration (Cmin) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Average Serum Concentration at steady state (Cav) | 0, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose
Accumulation Ratio (Rac) | 0, 0.5, 1, 2, 4, 8 hours post-dose on Day 1 and Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer